CLINICAL TRIAL: NCT01919151
Title: The Process of Metastasis in Colorectal Cancer Tumour Biology and Prognostic Factors in Pancreatic Cancer
Brief Title: Micrometastasis in Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 93-08172d6.2008.540
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Pancreatic Adenocarcinoma; Colorectal Cancer
Keywords: survival
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bone marrow cells fixated to slides or to cartridge. Some fresh frozen tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastrointestinal cancer patients: Patients with radiological suspected cancer in the pancreas Patients with radiological suspected colorectal liver metastasis

SUMMARY:
Prognostic and predictive value of assessing the patients micrometastasis status in blood and bone marrow when diagnosed GI cancer. 2 different patient subgroups are currently studied, patients with cancer of the pancreas and patients with liver metastasis secondary to colorectal cancer.

Our hypothesis is that patients with detective circulating tumor cells in the blood or disseminated tumour cells in their bone marrow at diagnosis have a more advanced disease than negative patients. This information may be of therapeutic interest.

DETAILED DESCRIPTION:
Oncological and overall outcome of the included patients are consecutively registrated at the out-patient clinic. At end of follow-up these survival data are analysed according to the presence of tumor cells in blood and bone marrow, and the prognostic impact of their presence are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven adenocarcinoma of the pancreas
2. Histological/radiological verified colorectal liver metastases
3. Consent capable patient
4. Signed written, informed consent

Exclusion Criteria:

1. Patient'history of other malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastrointestinal cancer patients:
  1. patients with suspected adenocarcinoma in the pancreas
  2. patients with liver metastases secondary to colorectal cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Atle Bjørnbeth, MD,PhD, Study Chair — Oslo University Hospital, Dep of Gastrointestinal surgery
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Hugenschmidt H, Labori KJ, Brunborg C, Verbeke CS, Seeberg LT, Bendigtsen Schirmer C, Renolen A, Borgen E, Naume B, Wiedswang G. Cytokeratin-positive cells in the bone marrow from patients with pancreatic, periampullary malignancy and benign pancreatic disease show no prognostic information. BMC Cancer. 2020 Nov 16;20(1):1107. doi: 10.1186/s12885-020-07510-z. PMID 33198661
- [Derived] Hugenschmidt H, Labori KJ, Brunborg C, Verbeke CS, Seeberg LT, Schirmer CB, Renolen A, Borgen EF, Naume B, Wiedswang G. Circulating Tumor Cells are an Independent Predictor of Shorter Survival in Patients Undergoing Resection for Pancreatic and Periampullary Adenocarcinoma. Ann Surg. 2020 Mar;271(3):549-558. doi: 10.1097/SLA.0000000000003035. PMID 30216219
- [Derived] Seeberg LT, Brunborg C, Waage A, Hugenschmidt H, Renolen A, Stav I, Bjornbeth BA, Borgen E, Naume B, Brudvik KW, Wiedswang G. Survival Impact of Primary Tumor Lymph Node Status and Circulating Tumor Cells in Patients with Colorectal Liver Metastases. Ann Surg Oncol. 2017 Aug;24(8):2113-2121. doi: 10.1245/s10434-017-5818-2. Epub 2017 Mar 3. PMID 28258416